CLINICAL TRIAL: NCT02071056
Title: Tissue and Fluid Collection Pilot Study to Develop Circulating Tumor DNA in Cerebrospinal Fluid as an Early Biomarker of LM in Patients With Metastatic Solid Tumor Cancer
Brief Title: Circulating Tumor DNA in Cerebrospinal Fluid as an Early Biomarker of Leptomeningeal Metastasis (LM)
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Lara K. Ronan, Assistant Professor Neuro-Oncology, Dartmouth-Hitchcock Medical Center
Other Study IDs: D13237
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Leptomeningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CSF and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- history of visceral cancer

SUMMARY:
The purpose of this study is to learn whether the DNA from cancer tumor cells can be found in the cerebral spinal fluid (CSF) that bathes the brain and spinal cord of patients before malignant the cancer cells themselves are able to be found in the CSF. The researchers doing this study hope this information can be used to develop a way to diagnose LM earlier .

DETAILED DESCRIPTION:
The contents of dead/dying tumor cells can be detected in the bloodstream, and this may be enhanced by the leaky vasculature of solid tumors. Circulating tumor DNA has been detected in plasma from patients with osteosarcoma, breast cancer, and colorectal cancer, and in cerebrospinal fluid from patients with cancer-associated neoplastic meningitis. Until recently, it was impractical to develop an assay to routinely quantify circulating tumor DNA due to heterogeneity between patients and tumors. Advances in genomic technology now permit sequencing a tumor genome to identify patient-specific genomic aberrations. Major genomic alterations (i.e., insertions, amplifications, deletions, inversions, translocations) can be readily detected using PCR primers and probes which will recognize tumor DNA but not normal DNA, permitting creation of a personalized assay to quantify tumor DNA levels in bodily fluids. We therefore propose a pilot study to determine whether circulating tumor DNA levels increase in CSF prior to cytological evidence of LM in patients with a history of cancer originating from a visceral organ.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a previously diagnosed solid tumor malignancy originating from a visceral organ (i.e., outside of the CNS), and present with signs and/or symptoms consistent with carcinomatous meningitis (headache, vision dysfunction, hearing loss, cranial nerve deficit, cognitive dysfunction, focal weakness or numbness suggestive of cranial neuropathy or radiculopathy, cauda equine syndrome, meningismus, and/or bowel or bladder dysfunction).
2. Age ≥ 18 years.
3. Patients will meet accepted standard of care and follow FDA guidance for low molecular weight heparin use prior to lumbar puncture, specifically INR < 1.4 and PT within normal range for DHMC laboratory, and platelet count >50,000. For enoxaparin use, delay of Lumbar puncture to allow at least 12 hours after administration of prophylactic doses, such as those used for prevention of deep vein thrombosis. Longer delays (24 hours) are appropriate to consider for patients receiving higher therapeutic doses of enoxaparin (1 mg/kg twice daily or 1.5 mg/kg once daily). A postprocedure dose of enoxaparin should usually be given no sooner than 4 hours after lumbar puncture. Aspirin and other antiplatelet therapy is permitted without timing constraints prior to or after lumbar puncture.
4. Patient must consent to provide up to additional CSF (10 mL) and blood (10 mL) when these fluids are drawn as part of clinically indicated procedures.
5. Patient must consent to permit genetic analysis of their cancer.
6. Patient capable of giving informed consent.
7. MRI of clinically symptomatic area (spine and/or brain) and/or head CT within the last 3 months to exclude brain disease that would contraindicate lumbar puncture.

Exclusion Criteria:

1. Evidence of a CNS mass creating mass-effect or midline shift such that lumbar puncture is contraindicated.
2. Previous or current hematological malignancy.
3. Previous or current primary CNS malignancy.
4. Prior treatment for CNS metastasis.
5. Known CNS autoimmune or inflammatory disease (i.e., Multiple Sclerosis, neurosarcoidosis, chronic fungal, rickettsial or bacterial meningitis).
6. Patient is currently receiving treatment for LM.
7. Patient was previously diagnosed with LM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurology and Medical Oncology clinical practices
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-11-25 (Actual); Study Completion 2015-11-25 (Actual)

PRIMARY OUTCOMES:
Tumor DNA detectability and cytological confirmation of leptomeningeal metastasis. | one year
  To determine whether circulating tumor DNA can be identified in the CSF of patients prior to cytological evidence of leptomeningeal metastasis in patients with a history of visceral cancer

SECONDARY OUTCOMES:
Comparison of circulating tumor DNA levels in CSF with levels in plasma. | one year
  To determine whether circulating tumor DNA levels in CSF correlate with levels in plasma.
Correlation of circulating tumor DNA levels and patient survival. | one year
  To determine whether circulating tumor DNA levels are predictive of patient survival.
Circulating tumor DNA detection in CSF of patients with cytological evidence of leptomeningeal metastasis. | one year
  To determine whether circulating tumor DNA is detectable in CSF of patients with cytological evidence of leptomeningeal metastasis.
Circulating tumor DNA identification in the CSF of patients prior to diagnosis of leptomeningeal metastasis. | one year
  To determine whether circulating tumor DNA can be identified in the CSF of patients prior to diagnosis of leptomeningeal metastasis.
Measurement of circulating tumor DNA levels and cancer cell numbers in CSF following initiation of intrathecal chemotherapy for leptomeningeal metastasis. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Lara K Ronan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States